CLINICAL TRIAL: NCT05878483
Title: Autonomous Blood Drawing Optimization and Performance Testing
Acronym: ADOPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vitestro B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL80965.000.22
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Venipuncture; Phlebotomy
Keywords: Autonomous; Blood Drawing; Phlebotomy; Robotics

STUDY DESIGN:
Intervention Model Description: Anticipated number of participants distribution:
  Phase A: 1,500 participants (max) Phase B1: 374 participants Phase B2/C1: 1,500 participants (max) Phase C2: 8,744 participants Phase 0: 1,500 participants (max)
  The Phases are sequential, reflective of technology development:
  Phase B1 should be completed before Phase B2/C1 can start. Phase B2 should be completed before Phase C2 can start.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autonomous blood drawing (Experimental): Hospital Sites (outpatients visiting blood drawing department):
  In study Phase A1, B1, B2, C1, a subject visiting the outpatient blood drawing department will receive one automated blood draw with the Venipuncture Device. This blood draw is additional to the manual blood draw.
  In study Phase C2 the automated blood draw replaces the manual blood draw. In Phase C2, the subject might therefore receive two automated blood draws, in case a redraw is required.
  Vitestro Site (volunteers):
  In study Phase A, C1 volunteers visit Vitestro Site. Participants receive one to two automated blood draws.
  Interventions: Device: Venipuncture Device (VD)

INTERVENTIONS:
Device: Venipuncture Device (VD) — The Venipuncture Device is a pre-market medical device that fully automates the blood drawing procedure (also called phlebotomy or venipuncture). It automatically detects a vein using near-infrared and ultrasound imaging technology, robotically inserts a needle, automatically connects blood tubes and applies pressure to the puncture site.
  During the ADOPT Study, the technology is further improved over time; for example features are released (such as: automated tourniquet). Initially, several manual steps are required to be performed by a device supervisor and operator. At the final stage of the ADOPT Study, Phase C2, the device has full functionality and only limited manual steps are required to be performed by a device supervisor.

SUMMARY:
The purpose of this pre-market clinical study is to evaluate the performance (efficacy) and safety of an autonomous blood drawing device (Venipuncture Device).

The study consists of several phases (A, B1, B2, C1, C2, 0).

Phase B1 is a confirmatory, Pivotal Clinical Study, required for regulatory approval, in which non-inferiority should be demonstrated in comparison to manual blood drawing.

Phases A, B2, C1, C2 are all exploratory studies, in which the technology and usability is further improved and tested. Phase 0 is an exploratory study for non-invasive technology testing (for example for improvement of ultrasound detection).

The study locations are outpatient blood drawing departments, in which patients are included as subjects. Additionally, in Phase A and C1, a small number of volunteers is included in a non-hospital site (Vitestro Site).

ELIGIBILITY:
Inclusion Criteria:

• Age ≥16 years.

Exclusion Criteria:

* Unable to follow instructions, due to mental disability and/or incapacity
* Unable to use device correctly due to physical impairment or disability (for example a patient with severe contractures or deformities)
* No venipuncture possible in cubital fossa of both arms (for example: after amputation of both arms)
* No venipuncture possible in cubital fossa due to contra-indications in both arms (for example: tattoos in both arms)
* Incapacitated persons
* Pregnant or breast-feeding

The following contra-indications / exclusion criteria are respected per arm:

* Arteriovenous fistula or vascular graft
* Paretic or paralyzed arm (e.g. after stroke or trauma)
* Infected skin in cubital fossa (for example: erysipelas or cellulitis)
* Mastectomy side, axillary lymph node excised
* Healed skin burns in cubital fossa
* Edema in cubital fossa
* Extensive scarring in cubital fossa
* Hematoma in cubital fossa
* Tattoos in cubital fossa

In case the test subject has a suitable contralateral arm, the subject can be included in this study. In Study Phase B2, a manual venipuncture and automated venipuncture are performed in both arms. Patients who have a contra-indication in one arm are excluded from the Phase B2 study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13618 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
First-time venipuncture success rate | Baseline
  Phase A/B1/B2/C1:
  Success is defined as blood flowing into blood tubes at first attempt; Failure is defined as no blood flowing in the blood tubes at all at first attempt.
  Phase C2: All blood tubes are filled sufficiently, no second venipuncture is required to obtain (all) the samples.

SECONDARY OUTCOMES:
Rate of punctured participants | Baseline
  The total number of participants that are punctured by the device is divided by the total number of included participants.
Rate of hemolyzed samples | Baseline
  All samples with an (automated) hemolysis-index of >0.5 hemoglobin g/l, are classified as hemolyzed. In the laboratories where reporting occurs in umol/l, 0.5 g/l is divided by a factor: 0.5 g/l / 1.6129= 31 umol/l.
Adverse Events | 7 days
  Number and type of Adverse Events (AE)s and Device Adverse Effects (ADEs) will be recorded and collected. A passive one week (7 days) follow-up occurs to determine whether any delayed adverse events occur.

CONTACTS AND LOCATIONS:
Overall Officials: Luuk Giesen, MD, Principal Investigator — Vitestro B.V.
Locations (5):
- Netherlands (5):
  - OLVG Lab, Amsterdam, North Holland
  - Amsterdam UMC, Amsterdam, North Holland
  - Result Laboratorium, location Albert Schweitzer Hospital, Dordrecht, South Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - Vitestro, Utrecht

IPD SHARING:
Plan to Share IPD: No